CLINICAL TRIAL: NCT02469623
Title: Dipole Density Right (and Left) Atrial Mapping and Assessment of Therapy In Complex Supraventricular Tachycardia
Brief Title: Dipole Density Mapping in Supraventricular Tachycardia
Acronym: DDRAMATIC-SVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-SVT-005; CL-SVT-002 (Other Grant/Funding Number: Acutus Medical); CL-SVT-001 (Other: Acutus Medical); CL-SVT-004 (Other: Acutus Medical); CL-SVT-006 (Other: Acutus Medical); CL-SVT-008 (Other: Acutus Medical); NCT01875614 (obsolete NCT alias); NCT01914549 (obsolete NCT alias); NCT01921660 (obsolete NCT alias); NCT02469636 (obsolete NCT alias); NCT02469649 (obsolete NCT alias)
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Dipole Density Mapping (Experimental)
  Interventions: Device: Dipole Density Mapping with AcQMap followed by ablation

INTERVENTIONS:
Device: Dipole Density Mapping with AcQMap followed by ablation

SUMMARY:
Use of dipole density mapping to identify activation in complex supraventricular tachycardias.

DETAILED DESCRIPTION:
The research study was conducted in multiple countries throughout the EU and Canada. The protocol and their corresponding NCT numbers are as follows:

NCT01914549 (Protocol CL-SVT-001, Site Belgium, Bruges Dr. Duytschaever = PI) NCT01875614 (Protocol CL-SVT-002, Sites in the UK, Drs. Grace, Hall, & Schilling = PIs) NCT03368781 (Protocol CL-SVT-004, Site Hamburg, Germany Prof. Willems = PI) NCT02469623 (Protocol CL-SVT-005, Site Prague, Czech Republic Prof. Neuzil = PI) NCT02469636 (Protocol CL-SVT-006, Site Santiago, Chile Dr. Bittner = PI) NCT02469649 (Protocol CL-SVT-008, Site Ontario, Canada Dr. Verma = PI)

All of the above records were combined into one as all protocols were essentially identical and one study report was written that encompasses the data/results for all protocols.

ELIGIBILITY:
Inclusion Criteria

1. Be aged 18-75 years
2. Be scheduled for ablation of an SVT due to the arrhythmia being recurrent, poorly tolerated, and /or unable to be controlled with antiarrhythmic drugs.
3. Be able and willing to give informed consent

Exclusion Criteria

1. Have any of the following:

   * implanted prosthetic, artificial, or repaired cardiac valves in the chamber being mapped
   * permanent pacemaker or ICD leads in the chamber being mapped
   * hypercoagulopathy or an inability to tolerate anticoagulation during the procedure
   * Stents in the area of the pulmonary veins (Study CL-SVT-004 ONLY)
2. MI within the prior two (2) months
3. Cardiac surgery within the prior three (3) months
4. Intracardiac thrombus
5. Clinically significant tricuspid and/or mitral valve regurgitation or stenosis
6. Cerebral ischemic event (including TIA) in the prior six (6) months
7. Pregnant or nursing
8. Currently enrolled in another clinical investigation
9. Have a contraindication for transfemoral venous access (Study CL-SVT-004 ONLY)
10. Have a contraindication for transseptal left atrial access (for patients with left atrial arrhythmias) (Study CL-SVT-004 ONLY)
11. Life expectancy of less than one (1) year (Study CL-SVT-004 ONLY)
12. Any health condition that, in the Investigator's opinion, would not allow the application of the investigational device (Study CL-AF-004 ONLY)

NOTE: The additional exclusion criteria for CL-SVT-004 were not expected to alter or bias the patient selection for study enrollment. While these criteria would have been assumed by other investigators as a standard of care for safe enrollment in a clinical study, the German EC approval required the additional statements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-09-06 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Nemocnice Na Homolce
Locations (8):
- AZ Sint-Jan AV Cardiologie, Bruges, Belgium
- Southlake Regional Health Center, Newmarket, Ontario, Canada
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Na Homolce Hospital, Prague, Czechia
- Elektrophysiologie Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- United Kingdom (3):
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Health NHS Trust, Whitechapel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grace A, Willems S, Meyer C, Verma A, Heck P, Zhu M, Shi X, Chou D, Dang L, Scharf C, Scharf G, Beatty G. High-resolution noncontact charge-density mapping of endocardial activation. JCI Insight. 2019 Mar 21;4(6):e126422. doi: 10.1172/jci.insight.126422. eCollection 2019 Mar 21. PMID 30895945

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Subjects: Subjects scheduled for an ablation of a supraventricular tachycardia due to the arrhythmia being recurrent using the AcQMap High Resolution Imaging and Mapping System (AcQMap System) in gathering data to create right and/or left atrial dipole density activation maps in subjects with supraventricular tachycardias (SVTs).
Period: Overall Study
Arm/Group | Treated Subjects
Started | 85
Completed | 72
Not Completed | 13
Not completed — Not consented for long-term follow-up | 4
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Groups:
- Dipole Density Mapping: Subjects scheduled for an ablation of a supraventricular tachycardia due to the arrhythmia being recurrent using the AcQMap High Resolution Imaging and Mapping System (AcQMap System) in gathering data to create right and/or left atrial dipole density activation maps in subjects with supraventricular tachycardias (SVTs).
  Follow-up is 7-10 days for non-AF patients (except in Germany where all subjects were followed for 1 year) and 1 year for AF patients following the procedure for each patient.
Arm/Group | Dipole Density Mapping
Number analyzed (Participants) | 85
Age, Continuous [Median (Standard Deviation); unit: years] | 59.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 85
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10
  Belgium | 2
  Czechia | 29
  United Kingdom | 29
  Chile | 3
  Germany | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Device-and Procedure-related Adverse Events and Serious Adverse Events
Description: Sites reported all adverse events throughout the study follow-up period regardless of their relationship to the device or procedure. Each event was classified and adjudicated by the site-specific investigator. The data were further analyzed by the Sponsor medical reviewer, providing a consistent determination of relationship to device, procedure and the subjects' underlying disease of the atrial arrhythmia condition.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Subjects
Number analyzed (Participants) | 85
Participants
  AF Subjects | 71
  Non-AF Subjects | 14
  Freedom a device related SAE @ 7dys | 85
  Freedom from a procedure-related SAE @ 7-dys | 83
  Freedom from an related AcQGuide SAE @ 7-dys | 71
  Freedom from a device related AE @ 7-days | 85
  Freedom from a procedure-related AE @ 7-days post | 64
  Freedom from an AcQGuide Sheath related AE @ 7-day | 71

2. Primary Outcome: The Number of Patients for Which Activation Maps Can be Created
Description: The primary performance endpoint was the number of subjects with successful construction of pre- and post-ablation procedure activation maps.
Time Frame: 1 day
Population: The study population consists of men and women between the ages of 18 - 75 years of age scheduled for an endocardial ablation for a supraventricular tachycardia (SVT)
Measure: Number; unit: participants
Groups:
- Subjects Scheduled for Ablation of an SVT: Subjects scheduled for ablation of a supraventricular tachycardia (SVT) due to the arrhythmia being recurrent, poorly tolerated and/or unable to be controlled with antiarrhythmic drug therapy
Arm/Group | Subjects Scheduled for Ablation of an SVT
Number analyzed (Participants) | 85
participants
  Pre-procedure activation maps | 83
  Post-procedure activation maps | 71

ADVERSE EVENTS:
Time Frame: Follow-up is 7-10 days for non-AF subjects (except in Germany where all subjects were followed for 1 year) and 1 year for AF patients following the procedure for each subject.
Arm/Group | Treated Subjects
All-Cause Mortality (participants affected / at risk) | 3/85
Serious Adverse Events (participants affected / at risk) | 10/85
Other Adverse Events (participants affected / at risk) | 30/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=85)
Access site Injury (Surgical and medical procedures) | 1 (1) — Hematoma right groin. Resolved without treatment. Remained in hospital for observation
Ablation re-do requiring hospitalization (Surgical and medical procedures) | 1 (1) — Atrial Fibrillation ablation Re-do
Valve Dysfunction (Surgical and medical procedures) | 1 (1) — Worsening of mitral valve regurgitation
Acute renal Insufficiency (Renal and urinary disorders) | 1 (1) — Patient was hospitalized due to acute renal insufficiency with anuria, hyperkalemia and signs of systemic infection of unknown etiology.
Carcinomamammae sin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Pt undergone the surgical resection on 18/NOV/2016 and was discharged from hospital on 22-Nov-2016. Recent check confirmed that marker tumors are normal.
Shortness of Breath (Cardiac disorders) | 1 (1) — Progressive shortness of breath secondary to noted heart failure
Arrhythmia (Cardiac disorders) | 1 (1) — On 09-MAY-2016 the pacemaker was implanted due to poly-arrhythmia symptoms and due to bradycardia.
Brain Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient was experiencing memory loss. The patient was assessed, CT head performed, followed by an MRI of the head. Diagnosis of glioblastoma multiforme
Death (Cardiac disorders) | 1 (1) — Cardiac Arrest
Abnormal Thyroid Function (Endocrine disorders) | 1 (1) — Post ablation admitted with abnormal thyroid function labs. Amiodarone stopped
Chest Infection (Infections and infestations) | 1 (1) — Patient thought to have developed chest infection. Antibiotics started and discharged 18 May 2016
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Patient went into fast AF rate 160, this lasted 3-4 hours. The event returned, and the patient was treated at another hospital and pacemaker was inserted on the 3rd August 2016
Atrial Flutter (Cardiac disorders) | 1 (1) — Patient presented to emergency room in flutter. He was given 500mcg x 2 Digoxin and this terminated the flutter into AF. He was discharged the following day.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=85)
Abnormal ECG (Cardiac disorders) | 1 (1) — Right bundle branch block
Abnormal lab value/infection (Infections and infestations) | 1 (1) — Leukocytosis as noted by changes in lab values. Controlled by primary care Doctor.
Access site injury (Surgical and medical procedures) | 14 (14) — groin hematoma
Atrial Fibrillation (Cardiac disorders) | 1 (1) — AF recurrence with dyspnea and fatigue
Air embolism/ST change (Surgical and medical procedures) | 1 (1) — An apparent air embolism from the AcQGuide Sheath caused a brief (1-2 min) change in ST segment that resolved without treatment
Arm Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Broken neck of the Humerus
Chest Pain (Cardiac disorders) | 1 (1) — Patient described retrosternal chest pain. Echocardiogram shows no pericardial effusion. Mild analgesics prescribed
Diarrhea (Gastrointestinal disorders) | 1 (1) — Rivaroxaban stopped - Apixaban started due to Diarrhea
Dizziness and Syncope (Cardiac disorders) | 1 (1) — Then patient complains of feeling frequently dizzy and as though he will pass out. ECG today shows sinus rhythm at 49bpm. No treatment prescribed
Exertional Dyspnea (Cardiac disorders) | 1 (1) — Dyspnea on Exertion. Sotolol discontinued
Groin Hematoma (Surgical and medical procedures) | 4 (4) — Groin Hematoma
Hemorrhoid Bleeding (Blood and lymphatic system disorders) | 1 (1) — Hemorrhage from Hemorrhoid
Hypertension (Cardiac disorders) | 2 (2) — Hypertension
Infection (Infections and infestations) | 1 (1) — Infection
Lower Extremity Swelling (General disorders) | 1 (1) — Swelling of Lower Extremities
Pericarditis (Cardiac disorders) | 1 (1) — Patient developed pericarditis 48 hr. post procedure, resolved with NSAIDS.
Pleuritic Chest pain (Cardiac disorders) | 1 (1) — Patient suffered pleuritic chest pain post procedure. Negative work up and mild analgesics prescribed.
Shortness of breath (Cardiac disorders) | 1 (1) — By 7 days FU, patient mentioned shortness of breath. Negative chest work up. Abnormal labs for thyroid function noted. AAD medication changed
Stumble/Fall (General disorders) | 1 (1) — Stumble fall on the street
Swollen Legs (General disorders) | 1 (1) — Swollen Legs. Amlodipine discontinued
Symptomatic Palpitations (Cardiac disorders) | 1 (1) — Palpitations and extra systolic beats
Syncope (Cardiac disorders) | 1 (1) — Syncopal episodes
Tonsilitis (Endocrine disorders) | 1 (1) — Tonsilitis
Vertigo (General disorders) | 1 (1) — Patient feels dizzy and had a hematoma in the right eye. 24 hours post-procedure diagnosed with recurrent AF

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT02469623/Prot_SAP_000.pdf